# STATISTICAL ANALYSIS PLAN Version 2.0

# EFFECTS OF FINGOLIMOD (GILENYA®) ON CYTOKINE AND CHEMOKINE LEVELS IN RELAPSING REMITTING MULTIPLE SCLEROSIS PATIENTS

STUDY NUMBER: FTY720/Fingolimod

STUDY NAME: BIYOMARKER

# Statistical Analysis Plan Signature Page

# Version 2.0

| Sponsor | : | NOVARTIS | |
|---|---|---|---|
| Protocol | : | [CFTY720DTR04] / NCT02373098 | |
| Study title | : | _ | on Cytokine and Chemokine<br>Itiple Sclerosis Patients |
| | , Bio., N | I.Sc. | 30.11.2017 |
| Author | | | Date |
| Reviewed by | | | Date |
| | , M.D. | | 04.12.2017 |
| Approved by | | | Date |

# TABLE OF CONTENTS

| 1 | ABBREV | VIATIONS | 4 |
|------|--------|-------------------------------------------|---|
| 2 | BACKGF | ROUND | 5 |
| 3 | OBJECT | IVES OF THE STUDY | 5 |
| 3.1. | Prima | ıry Objective | 5 |
| 3.2. | Secon | dary Objective | 5 |
| 4 | | DESIGN | |
| 5 | ANALYZ | ED POPULATIONS | 7 |
| 5.1. | | le Size Calculation | |
| 6 | | SIS PLAN | |
| 6. | | nographics | |
| 6. | | NICAL DATA | |
| 6. | | BORATORY TESTS | |
| | 6.3.1 | Clinical Biochemistry | |
| | 6.3.2 | Hematology | |
| 6. | | SESSMENTS OF SCALE | |
| 6. | | SESSMENT OF CYTOKINE AND CHEMOKINE LEVELS | |
| 0. | 6.5.1 | ELISA | |
| | 6.5.1 | | |
| , | | Flow Cytometry | |
| 6. | U SAI | FETY ASSESSMENT | Y |

### 1 ABBREVIATIONS

AE Adverse Event

ALT Alanine aminotransferase

AST Aspartate aminotransferase

CCL2 Chemokine (C-C motif) ligand 2

CXCL13 Chemokine (C-X-C motif) ligand 13

CXCR3 Chemokine (C-X-C motif) receptor 3

ELISA Enzyme-linked Immunosorbent Assay

EDSS Expanded Disability Status Scale

GCP Good Clinical Practice

ICH International Conference on Harmonisation of Technical Requirements for

Registration of Pharmaceuticals for Human Use

MS Multiple Sclerosis

PASAT Paced Auditory Serial Addition Test

RRMS Relapsing-remitting Multiple Sclerosis

SAE Serious Adverse Event

SDMT Symbol Digit Modalities Test

TNF Tumor Necrosis Factor

VLA Very Late Antigen

WBC White Blood Cell

#### 2 BACKGROUND

The purpose of this statistical plan is to define the tables, lists, data summaries and graphs to be prepared and to determine the statistical methods to be used for the analysis of the results of the study titled, "Effects of Fingolimod (Gilenya®) on Cytokine and Chemokine Levels in Relapsing Remitting Multiple Sclerosis Patients".

This statistical analysis plan has been prepared in pursuant to and in line with ICH-GCP principles and protocol no. CFTY720DTR04.

## **3 OBJECTIVES OF THE STUDY**

#### 3.1. PRIMARY OBJECTIVE

The primary objective of this study is to evaluate the differences between serum cytokine and chemokine levels of healthy controls and multiple sclerosis patients.

## 3.2. SECONDARY OBJECTIVE

The secondary objective of this study is to test the predictive value of cytokine/chemokine changes measured in the 3rd and 6th months on the PASAT, SDMT, 9-Hole peg test, timed 25-foot walk, EDSS and relapse rate observed after 6 months of treatment.

# 4 STUDY DESIGN

This study is a multi center, open label study.

80 relapsing remitting MS (RRMS) patients will be recruited according to the Mc Donald's criteria and 60 healthy controls will be recruited as the control group. All subjects will sign an informed consent that will be approved by the local Ethics Committee and the applicable health authorities prior to venipuncture. Basal EDSS, relapses during the last 2 years, paced auditory serial addition task (PASAT), 9-Hole peg test, timed 25-foot walk and single digit modalities test (SDMT) scores will be recorded before study entry. Serum and blood samples will be collected from each participant after evaluation for inclusion and exclusion criteria. Additional serum and blood samples at 2 different time points will be collected from MS patients at months 3 (±1 week) and 6 (±2 weeks) after starting fingolimod 0.5 mg/day po. treatment (Figure 1). Serum samples will be stored at -20oC at local centers for a longest duration of two weeks and kept frozen at -80°C

until assayed. The levels of IL-4, IL-6, IL-8, IL-9, IL-10,

IL-13, IL-17, IL-23, IFN-γ, TNF-α, VLA4, CCL2, CCL5, CXCR3, CXCL13 will be measured by ELISA according to the manufacturer's protocols. Optical density (OD) will be measured at 450 nm and cytokine/chemokine concentrations (pg/ml) will be calculated by referring to a standard curve.

Whole blood samples will be dispatched

In order to perform flow cytometry assay for intracellular cytokine measurement PBMC will be isolated freshly.

EDSS and relapses will be recorded after 6 months of treatment. PASAT, 9-hole peg test, timed 25-foot walk and SDMT's will be performed only at study entry and termination after 6 months (Figure 1).

**Figure 1:** Study protocol (PASAT: Paced auditory serial addition task, SDMT: single digit modalities test, FACS: Flow assisted cell sorting, flow cytometry)



### 5 ANALYZED POPULATIONS

The study will include only 80 relapsing remitting MS patients and 60 healthy controls without any known autoimmune disease. RRMS patients will be followed for 6 months.

# 5.1. SAMPLE SIZE CALCULATION

Due to the lack of previous studies using all of the cytokines and chemokines and multitudinous analyses, it is difficult to estimate a precise sample size for our study. Despite this, our previous publications indicate that the basal IL-17 concentration is normally distributed with a mean of 32 pg/ml (±stdev of 15 pg/ml) in RRMS patients. If the true difference in the mean concentration of matched pairs is 7 pg/ml, we will need to study 50 pairs of subjects to be able to reject the null hypothesis with a power of 90%. The Type I error probability associated with this test of this null hypothesis is 0,05.

With assumption of drop out rate of 20% minimum 60 RRMS patients and 60 healthy control subjects should enroll to the study. Due to expected high rate of screen failure patients, we decided to screen 80 RRMS patients in order to reach 60 eligible RRMS subjects for the study.

# 6 ANALYSIS PLAN

Data analysis will be performed after all of the data is collected from the enrolled patients. All MS patients and control group will be accepted as the analysis sets.

Cytokine and chemokine levels will be analyzed cumulatively at the end of the study. The results will be recorded to the blood sampling logs and laboratory logs cumulatively.

### 6.1 DEMOGRAPHICS

- Gender: Subjects, male and female, in both groups (Control & MS patients) will be expressed separately as n and %.
- Age: Age data for subjects in the "Control" and in the "MS patients" groups will be tabulated by calculating n, mean, standard deviation, minimum, maximum and median.

Page 7/9

# 6.2 CLINICAL DATA

- **Previous MS treatment** of the patients will be expressed as n and %.
- Age of onset of MS of the patients will be tabulated by calculating n, mean, standard deviation, minimum, maximum and median.
- **Duration of MS (years)** of the patients will be tabulated by calculating n, mean, standard deviation, minimum, maximum and median.
- MS relapses in the previous 2 years of the patients will be tabulated by calculating n, mean, standard deviation, minimum, maximum and median.
- MS relapses requiring corticosteroids in the previous 2 years of the patients will be tabulated by calculating n, mean, standard deviation, minimum, maximum and median.
- MS relapses in the previous 1 year of the patients will be tabulated by calculating n, mean, standard deviation, minimum, maximum and median.
- MS relapses requiring corticosteroids in the previous 1 year of the patients will be tabulated by calculating n, mean, standard deviation, minimum, maximum and median.
- **Duration of treatments (months)** of the patients will be tabulated by calculating n, mean, standard deviation, minimum, maximum and median.
- Relapse rates of the patients will be evaluated.

### 6.3 LABORATORY TESTS

# 6.3.1 Clinical Biochemistry

Patients' AST, ALT, BUN, Creatinine, Total Cholesterol, Tryglicerides, LDL-C, HDL-C, TSH, ST4, Glucose and HbA1c values will be tabulated by calculating mean and standart deviation and compared as Visit 1 vs. Visit 2 and Visit 1 vs. Visit 3 by using appropriate statistical test. Wilcoxon test will be used in the dependent variables with non-normal distributions whereas Paired sample t test will be used in the dependent variables with normal distributions.

## 6.3.2 Hematology

Patients' WBC, Absolute Lymphocyte Count, Platelet, Absolute Neutrophil Count and Hemoglobin values will be tabulated by calculating mean and standart deviation and compared as Visit 1 vs. Visit 2 and Visit 1 vs. Visit 3 by using appropriate statistical test. Wilcoxon test will be used in the dependent variables with non-normal distributions whereas Paired sample t test will be used in the dependent variables with normal distributions.

#### 6.4 ASSESSMENTS OF SCALE

Patients' EDSS, PASAT, SDMT, 9-hole peg test and timed 25-foot walk test values will be tabulated by calculating mean and standart deviation and compared as Visit 1 vs. Visit 3 by using appropriate statistical test. Wilcoxon test will be used in the dependent variables with non-normal distributions whereas Paired sample t test will be used in the dependent variables with normal distributions.

### 6.5 ASSESSMENT OF CYTOKINE AND CHEMOKINE LEVELS

#### **6.5.1** ELISA

Subjects' IL-4, IL-6, IL-8, IL-9, IL-10, IL-13, IL-17, IL-23, IFN-γ, TNF-α, VLA4, CCL2, CCL5, CXCR3 and CXCL13 values will be tabulated by calculating mean and standart error and compared as Control group vs. Visit 1 (MS patients), Visit 1 (MS patients) vs. Visit 2 (MS patients), Visit 1 (MS patients) vs. Visit 3 (MS patients) and Control group vs. Visit 3 (MS patients) by using appropriate statistical test. Mann Whitney U test with significance level of 0.05 was used for the independent variables since non-normal distributions had been observed. Wilcoxon test was used for the dependent variables with non-normal distributions. For the independent variables with normal distributions Independent Sample t test was used whereas Paired sample t test was used for the dependent variables with normal distributions.

# 6.5.2 Flow Cytometry

Subjects' IL-4, IL-6, IL-9, IL-10, IL-13, IL-17, IFN-γ and TNF-α values will be tabulated by calculating mean and standart error and compared as Control group vs. Visit 1 (MS patients), Visit 1 (MS patients) vs. Visit 2 (MS patients), Visit 1 (MS patients) vs. Visit 3 (MS patients) and Control group vs. Visit 3 (MS patients) by using appropriate statistical test. Mann Whitney U test with significance level of 0.05 was used for the independent variables since non-normal distributions had been observed. Wilcoxon test was used for the dependent variables with normal distributions. For the independent variables with normal distributions Independent Sample t test was used whereas Paired sample t test was used for the dependent variables with normal distributions.

## 6.6 SAFETY ASSESSMENT

Incidence of AEs, incidence of SAEs and number of patients who died or experienced other serious or clinically significant events will be tabulated.